CLINICAL TRIAL: NCT06777186
Title: Evaluation of Motor Skills, Balance, Dual Task, and Social Adaptation in Individuals with Autism
Status: Recruiting | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Simay Tepik, Physiotherapist, MASTER'S STUDENT, Kırıkkale University
Other Study IDs: Gurbuz07
Record Dates: First submitted 2025-01-10; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Autism Spectrum Disorder; Motor Disorders; Social Skills
MeSH Terms: conditions — Autism Spectrum Disorder; Motor Disorders; Social Skills

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Autism Spectrum Disorder
  Interventions: Other: 10 meter walk test; Other: Functional Balance; Other: Social Adaptation Assessment; Other: Motor skills and proficiency
- Healthy Children
  Interventions: Other: 10 meter walk test; Other: Functional Balance; Other: Social Adaptation Assessment; Other: Motor skills and proficiency

INTERVENTIONS:
Other: 10 meter walk test — The dual task skills of the individuals will be evaluated by adding motor and cognitive tasks to the 10-meter walk test. Tasks given to individuals
  Single motor task (comfortable walking): The individual is asked to walk at normal speed, the time is recorded Motor-motor dual task: Both hands carry a half-full water bottle, time is recorded Motor-cognitive dual task (mental) : counts backwards from 10 by 1, time is recorded Motor - cognitive dual task (memory) : The individual is asked to say 3 words that were previously spoken. The time is recorded.
Other: Functional Balance — It will be assessed with the TUG test. The TUG measures the time it takes for an individual to get up from a chair, walk a distance of 3 meters, turn around, walk back to the chair and sit down again after a ready, go signal.
Other: Social Adaptation Assessment — Adaptive behavior will be assessed with the Vineland Adaptive Behavior Scales. It is a parent interview designed to assess functioning in daily life. [35]Specifically, adaptive behavior is assessed in four domains: Communication, Daily Living, Socialization and Motor skills. Vineland has reliability and current validity. It has been reported to be sensitive to the difficulties experienced by children with ASD
Other: Motor skills and proficiency — The Bruininks-Oseretsky Motor Proficiency Test (BOT-2) assesses fine motor, hand coordination, body coordination, strength and agility between the ages of 4-21 years.There are 53 items in the BOT-2. In BOT-2, there are four motor domains including fine motor control, hand coordination, body coordination, strength and agility and a total of eight subtests related to these domains.

SUMMARY:
The aim of our study is to evaluate motor skills balance, dual task and social adaptation skills in individuals with autism. Our study will be conducted in Bartın Lider Special Education and Rehabilitation Center after ethics committee approval. The sample number determined by power analysis will be included in the study. Socio-demographic characteristics (age, height, body weight, body mass index, education level, exercise and smoking habits, etc.) of the individuals who voluntarily participated in the study will be obtained. The individuals participating in the study will be divided into two groups as individuals with normal motor development and individuals with autism spectrum disorder and the same assessment scales will be used. These assessment scales are TUG, 10 meter walking test, Vineland Adaptive Adaptation Scale, Bruininks-Oseretsky Motor Competence Test. According to the evaluation results, motor skills, functional balance, dual task and social adaptation skills of individuals with autism will be compared with individuals with normal motor development.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with ASD by a physician
* Children are receiving education in a special education and rehabilitation center
* No vision problems
* Ability to receive and execute commands
* No cognitive problems
* No walking problems

Exclusion Criteria:

* Individuals with concomitant secondary diseases
* Individuals who have undergone surgery in the last six months

Ages: 4 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: G*Power (version 3.1.9.4) package program was used for power analysis. Assuming that the effect size that could be obtained between the two groups would be large (f = 0.543 (EFFECT SIZE)), as a result of the power analysis, it was calculated that 80% power could be obtained at 90% confidence level (with a margin of error of 0.05) when at least 110 people were included in the study
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
10 meter walk test | At enrollment
  The dual task skills of the individuals will be evaluated by adding motor and cognitive tasks to the 10-meter walk test.

SECONDARY OUTCOMES:
Functional Balance | At enrollment
  It will be assessed with the TUG test. The TUG measures the time it takes for an individual to get up from a chair, walk a distance of 3 meters, turn around, walk back to the chair and sit down again after a ready, go signal.
Social Adaptation Assessment | At enrollment
  Adaptive behavior will be assessed with the Vineland Adaptive Behavior Scales. It is a parent interview designed to assess functioning in daily life. [35]Specifically, adaptive behavior is assessed in four domains: Communication, Daily Living, Socialization and Motor skills. Vineland has reliability and current validity. It has been reported to be sensitive to the difficulties experienced by children with ASD
Motor skills and proficiency | At enrollment
  The Bruininks-Oseretsky Motor Proficiency Test (BOT-2) assesses fine motor, hand coordination, body coordination, strength and agility between the ages of 4-21 years[37] There are 53 items in the BOT-2. In BOT-2, there are four motor domains including fine motor control, hand coordination, body coordination, strength and agility and a total of eight subtests related to these domains. The highest score to be obtained from this 53-item test is 320. A short form of this test with 14 items was created, and then it was reorganized in 2010 by reducing the number of items to 12. The highest score to be obtained during the application of the test is 72.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırıkkale University, Kırıkkale, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No